CLINICAL TRIAL: NCT02163213
Title: An Open-Label Study Evaluating the Impact of Serum-Derived Bovine Immunoglobulin /Protein Isolate (SBI) 5.0 g Twice Daily on Nutritional Status in Subjects With Diarrhea-Predominant Irritable Bowel Syndrome (IBS-D)
Brief Title: Serum-Derived Bovine Immunoglobulin /Protein Isolate (SBI) 5.0 g Bid on Nutritional Status in Subjects With IBS-D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Michael Camilleri, M.D., Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 14-002151
Record Dates: First submitted 2014-06-09; First posted 2014-06-13 (Estimated); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Diarrhea-predominant Irritable Bowel Syndrome
Keywords: diarrhea; irritable bowel syndrome
MeSH Terms: conditions — Diarrhea; Irritable Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Serum Bovine Immunoglobulin (Other): Serum-Derived Bovine Immunoglobulin (SBI) 5.0 g by mouth twice daily;
  Effects of SBI will be compared with observations and measurements performed at baseline PRIOR to starting the SBI treatment
  Interventions: Other: Serum-derived bovine immunoglobulin protein isolate (SBI)

INTERVENTIONS:
Other: Serum-derived bovine immunoglobulin protein isolate (SBI) — Serum-Derived Bovine Immunoglobulin /Protein Isolate (SBI) 5.0 g bid on Nutritional Status and intestinal functions in Subjects with IBS-D

SUMMARY:
To evaluate the safety and effectiveness of oral nutritional therapy Serum-Derived Bovine Immunoglobulin (SBI) on nutritional status, epithelial barrier function, and mucosal expression of pivotal genes including tight junction, secretory mechanisms, tissue repair proteins and chemokines in subjects with IBS-D.

DETAILED DESCRIPTION:
This is an open label study evaluating the impact of SBI 5.0 g twice daily on

1. nutritional status (plasma amino acid profile and kynurenine to tryptophan ratio),
2. intestinal permeability (in vivo) and
3. mucosal expression of pivotal genes including tight junction, secretory mechanisms, tissue repair proteins and chemokines status in patients with IBS-D.

Plasma, duodenal and stool samples will be collected. Fifteen eligible subjects will be enrolled to receive SBI for 8 weeks (SBI 5.0g BID for 8 weeks).

Intestinal permeability will be measured in vivo by two sugar urine excretion(s) after oral ingestion.

Biopsies from the distal second or third portion of the duodenum will be obtained endoscopically, to measure mRNA expression of tight junction proteins and markers of immune function,

ELIGIBILITY:
Inclusion criteria:

1. Age 18-65y
2. Male or non-pregnant female
3. IBS by Rome III criteria with predominant symptom of diarrhea
4. Baseline 14 day diary showing average of 2 days per week with >3 bowel movements per day

Exclusion criteria:

1. Intake of medications that interfere with the study
2. Antibiotic within prior 2 weeks and throughout study
3. Prior abdominal surgery except appendectomy
4. Active gastrointestinal diagnosis other than IBS
5. History of allergy or intolerance to beef or to any ingredient in the investigational product
6. Uncontrolled psychiatric disorders (includes significant depression or suicidal ideation), in investigator's judgment
7. Use of tobacco products within the past six months or nonsteroidal antiinflammatory drugs or aspirin within the past week (since they all may affect intestinal permeability)
8. Bleeding disorders or medications that increase risk of bleeding from mucosal biopsies.
9. For two days prior to studies, patients are instructed to avoid ingestion of artificial sweeteners such as Splenda trademark (TM) (sucralose), Nutrasweet TM (aspartame), foods containing lactulose or mannitol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-06; Primary Completion 2016-11-01 (Actual); Study Completion 2016-11-02 (Actual)

PRIMARY OUTCOMES:
Change in epithelial barrier function, and mucosal expression of barrier-associated genes | 10 weeks
  The primary endpoints for the study are change from baseline in mucosal expression of tight junction proteins (ZO-1, occludin, claudin)

SECONDARY OUTCOMES:
Change in body measurements, amino acid metabolism, abdominal pain, and baseline stool frequency and consistency. | 10 weeks
  The secondary endpoints for the study is change from baseline in amino acid metabolism

OTHER OUTCOMES:
Duodenal and fecal microbiomes | 10 weeks
  Exploratory endpoints: Duodenal biopsy microbiome

CONTACTS AND LOCATIONS:
Overall Officials: Michael Camilleri, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Wang XJ, Carlson P, Chedid V, Maselli DB, Taylor AL, McKinzie S, Camilleri M. Differential mRNA Expression in Ileal Mucosal Biopsies of Patients With Diarrhea- or Constipation-Predominant Irritable Bowel Syndrome. Clin Transl Gastroenterol. 2021 Apr 12;12(4):e00329. doi: 10.14309/ctg.0000000000000329. PMID 33843785